CLINICAL TRIAL: NCT07237308
Title: A Multicenter Prospective Randomized Study to Evaluate the Efficacy of Apixaban and Clopidogrel on the Prevention of Recurrent Ischemic Stroke in Patients With Atrial Fibrillation and Cerebral Atherosclerosis
Brief Title: BEACON-AA: Apixaban With or Without Clopidogrel in Stroke Patients With Atrial Fibrillation and Cerebral Atherosclerosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2025-0697
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Ischemic; Atrial Fibrillation; Intracrnaial Arterioscelrosis; Arteriosclerosis
MeSH Terms: conditions — Stroke; Ischemia; Atrial Fibrillation; Arteriosclerosis | interventions — apixaban; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban and Clopidogrel Combination Therapy (Experimental): Participants receive apixaban (5 mg or 2.5 mg if indicated) plus clopidogrel 75 mg daily for 30 days, followed by apixaban monotherapy thereafter.
  Interventions: Drug: Apixaban
- Apixaban Monotherapy (Experimental): Participants receive apixaban 5 mg (or 2.5 mg if indicated) once daily as monotherapy for 30 days and continue apixaban monotherapy thereafter.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Apixaban — Apixaban 5mg (or 2.5mg if indicated) once daily. Used as monotherapy or in combination with clopidogrel for 30 days, then continued as monotherapy.
  Other Names: Eliquis
  Arms: Apixaban and Clopidogrel Combination Therapy
Drug: Clopidogrel — Clopidogrel 75mg once daily for 30 days in combination with apixaban, then discontinued.
  Other Names: Plavix
  Arms: Apixaban Monotherapy

SUMMARY:
This trial aims to compare the safety and efficacy of apixaban alone versus apixaban combined with clopidogrel in patients with acute ischemic stroke associated with non-valvular atrial fibrillation and concomitant symptomatic intracranial or extracranial atherosclerosis. Participants will be randomly assigned in a 1:1 ratio to receive apixaban monotherapy or dual therapy with clopidogrel for 30 days. The primary outcome is the incidence of symptomatic or asymptomatic recurrent ischemic lesions detected on brain MRI (DWI/FLAIR) at 30 ± 5 days after initiation of study medication.

DETAILED DESCRIPTION:
"Although oral anticoagulants are effective in preventing cardioembolic stroke in patients with non-valvular atrial fibrillation (NVAF), a considerable proportion of ischemic strokes in these patients are caused by concomitant large artery atherosclerosis. Carotid or intracranial artery stenosis is present in a substantial number of patients with NVAF and is associated with a higher risk of recurrent cerebral infarction despite standard anticoagulation. In such patients, adding an antiplatelet agent to oral anticoagulation may theoretically reduce atherothrombotic events, but it also raises concern for increased bleeding risk. Recent clinical evidence on this issue remains limited, and the optimal antithrombotic strategy for patients with NVAF and coexisting symptomatic atherosclerotic stenosis has not been clearly established.

The BEACON-AA trial is a multicenter, randomized, open-label, blinded-endpoint (PROBE) study designed to compare the safety and efficacy of apixaban monotherapy versus apixaban combined with clopidogrel in patients with acute ischemic stroke associated with non-valvular atrial fibrillation (NVAF) and concomitant symptomatic intracranial or extracranial atherosclerosis. Participants will be randomized in a 1:1 ratio to receive apixaban alone or apixaban plus clopidogrel for 30 days, followed by apixaban monotherapy thereafter.

Brain MRI including diffusion-weighted and FLAIR sequences will be performed at baseline and at 30 ± 5 days to assess new or recurrent ischemic lesions. The primary efficacy outcome is the incidence of symptomatic or asymptomatic recurrent ischemic lesions detected on brain MRI (DWI/FLAIR) at 30 ± 5 days after initiation of study medication. Secondary efficacy outcomes include: 1) incidence of symptomatic ischemic stroke or transient ischemic attack within 90 days, 2) incidence of acute coronary syndrome within 90 days,3) cardiovascular mortality within 90 days, 4) composite major cardiovascular events within 90 days, 5) all-cause mortality within 90 days, 6) proportion of patients with modified Rankin Scale (mRS) 0-2 at 90 days, and 7) proportion of patients with mRS 0-3 at 90 days. The primary safety outcomes are: 1) incidence of major bleeding within 90 days, defined according to the International Society on Thrombosis and Haemostasis (ISTH) criteria and 2) incidence of new asymptomatic cerebral hemorrhages detected on brain MRI (DWI/FLAIR) at 30 ± 5 days after initiation of study medication. All imaging and clinical events will be independently adjudicated by blinded central adjudication committees."

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older at the time of enrollment.
2. Patients with non-valvular atrial fibrillation (NVAF) documented by electrocardiography or medical records.
3. Acute ischemic stroke confirmed by brain MRI (diffusion-weighted and FLAIR sequences), with neurological symptoms occurring within 5 days prior to randomization.
4. Presence of clinically significant atherosclerosis in the cerebral or aortic arteries, meeting at least one of the following criteria:

   ① ≥30% stenosis in the relevant artery (the artery supplying the infarcted territory) demonstrated by CTA, MRA, or DSA - using the WASID criteria for intracranial arteries and NASCET criteria for extracranial arteries.

   ② High-risk atherosclerotic plaque features in the relevant artery demonstrated by CTA, MRA, or ultrasound, such as ulceration, intraplaque hemorrhage, mobile plaque, or a large lipid core (involving ≥25% of plaque cross-sectional area) on CTA/MRA, or ulceration, mobile plaque, or hypoechoic/echolucent plaque on ultrasound; or presence of branch artery occlusive disease (BAOD).

   ③ Complex aortic plaque (≥4 mm in thickness, mobile, or ulcerative) identified in the ascending aorta or aortic arch by transthoracic/transesophageal echocardiography or coronary CT angiography.
5. Ability and willingness to provide written informed consent for participation in the study.

Exclusion Criteria:

1. Presence of mechanical heart valves or rheumatic mitral stenosis.
2. Requirement for antiplatelet agents other than clopidogrel.
3. Planned percutaneous coronary intervention, coronary artery bypass graft surgery, carotid endarterectomy, or intracranial stenting within 3 months after enrollment.
4. Presence of mural thrombus in the heart confirmed by imaging.
5. Renal impairment with creatinine clearance ≤30 mL/min/1.73 m².
6. Severe hepatic impairment, including acute hepatitis, chronic active hepatitis, hepatic lesions or coagulopathy, hepatic failure, or laboratory evidence of AST/ALT >2× the upper limit of normal (ULN) or total bilirubin >1.5× ULN.
7. Small-vessel occlusion (lacunar infarction) according to the TOAST classification.
8. History within the past 30 days of gastrointestinal bleeding, vascular malformation of the brain or spinal cord, recent brain, spinal, or ophthalmologic surgery or trauma, esophageal varices, or intracranial hemorrhage at any time; or chronic regular use of NSAIDs (≥3 days per week for ≥2 consecutive weeks).
9. Ischemic stroke occurring despite concurrent use of both NOAC and antiplatelet therapy.
10. Planned surgery or high-bleeding-risk procedure within 3 months, or presence of active bleeding at enrollment.
11. Anemia (hemoglobin < 8.0 g/dL) or thrombocytopenia (platelet count < 100,000/µL).
12. Pre-stroke modified Rankin Scale (mRS) ≥ 2.
13. Severe comorbid illness or malignancy not in complete remission with an expected life expectancy <1 year.
14. Known hypersensitivity or allergy to apixaban or clopidogrel.
15. Pregnant or breastfeeding women.
16. Uncontrolled diabetes mellitus (HbA1c > 10.0%) or severe hypertension (systolic ≥ 220 mmHg or diastolic ≥ 120 mmHg).
17. Concomitant use of strong CYP3A4 and P-glycoprotein inhibitors that can significantly increase apixaban exposure (e.g., ketoconazole, itraconazole, ritonavir, clarithromycin).
18. Concomitant use of strong CYP2C19 inducers that can reduce clopidogrel antiplatelet effect (e.g., rifampin, carbamazepine, phenytoin, phenobarbital, St. John's wort).
19. Clinically significant mass effect due to space-occupying cerebral infarction, or patients expected to require decompressive craniectomy, including those with midline shift > 5 mm, loss of basal cisterns, herniation, fourth-ventricle compression, or obstructive hydrocephalus in posterior fossa infarcts.
20. Intracranial hemorrhage or hemorrhagic transformation (PH1 or PH2) according to ECASS criteria.
21. Participation in another interventional clinical trial within the past 30 days or concurrent participation in another interventional study (non-interventional observational or registry studies may be allowed at the investigator's discretion).
22. Any other condition that, in the investigator's judgment, would make participation or continued involvement in the study inappropriate or infeasible.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic or asymptomatic recurrent ischemic lesions detected on brain MRI (DWI/FLAIR) | At 30 ± 5 days after initiation of study medication
  Recurrent ischemic lesions, either symptomatic or asymptomatic, identified on diffusion-weighted imaging (DWI) and FLAIR MRI performed at 30 ± 5 days following randomization.

SECONDARY OUTCOMES:
Incidence of symptomatic ischemic stroke or transient ischemic attack (TIA) | Within 90 days after randomization
  Occurrence of new symptomatic ischemic stroke or transient ischemic attack confirmed by clinical and/or imaging criteria.
Incidence of acute coronary syndrome (ACS) | Within 90 days after randomization
  Occurrence of acute coronary syndrome, including unstable angina or myocardial infarction, confirmed by standard diagnostic criteria.
Cardiovascular mortality | Within 90 days after randomization
  Death attributable to cardiovascular causes, including ischemic stroke, myocardial infarction, heart failure, or sudden cardiac death.
Composite major cardiovascular events | Within 90 days after randomization
  Composite of ischemic stroke/TIA, acute coronary syndrome, or cardiovascular death.
All-cause mortality | Within 90 days after randomization
  Death from any cause during the 90-day follow-up period.
Proportion of patients with modified Rankin Scale (mRS) score 0-2 | At 90 days after randomization
  Functional independence defined as mRS score of 0-2 at day 90.
Proportion of patients with modified Rankin Scale (mRS) score 0-3 | At 90 days after randomization
  Favorable functional outcome defined as mRS score of 0-3 at day 90.
Incidence of major bleeding events according to the ISTH criteria | Within 90 days after randomization
  Major bleeding events defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria, including fatal bleeding, symptomatic intracranial hemorrhage, intraocular bleeding causing vision loss, bleeding resulting in inability to perform usual activities, bleeding requiring transfusion of ≥2 units of whole blood or red cells, or bleeding leading to hospitalization.
Incidence of new asymptomatic cerebral hemorrhages detected on brain MRI (DWI/FLAIR) | At 30 ± 5 days after randomization
  Newly developed asymptomatic cerebral hemorrhages identified on diffusion-weighted and FLAIR MRI performed 30 ± 5 days after randomization.

IPD SHARING:
Plan to Share IPD: Undecided